CLINICAL TRIAL: NCT03713580
Title: A Phase I Trial of Venetoclax in Combination With BEAM Conditioning Regimen for Autologous Stem Cell Transplantation in Patients With Relapsed or Refractory Non-Hodgkin Lymphoma
Brief Title: Venetoclax in Combination With BEAM Conditioning Regimen for ASCT in Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2418
Record Dates: First submitted 2018-10-05; First posted 2018-10-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Non-hodgkin Lymphoma
Keywords: Autologous stem cell transplant (ASCT); Venetoclax
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Venetoclax+BEAM x 1 cycle prior to ASCT (Experimental): Venetoclax dose escalation cohorts + BEAM (Carmustine, Etoposide, Cytarabine, Melphalan) begin with dose level 1 (800mg on Day -7 and Day -6). The dosing cohorts are escalated in a 3 + 3 design but with increasing duration instead of increasing dosage.
  Carmustine 300 mg/m2 by IV over 2 hours on Day -7.
  Etoposide 100 mg/m2 by IV over 6 hours daily for 4 consecutive days, Day-6 through Day-3.
  Cytarabine 200 mg/m2 by IV over 2 hours every 12 hours for 3 consecutive days, Day-6 through Day-4.
  Melphalan 140 mg/m2 by IV over 30 minutes or IV push once on Day -2.
  Following V+BEAM therapy, participants will receive Autologous Stem Cell Transplant (ASCT): infusion of previously collected autologous stem cells and supportive care per institutional guidelines
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Adding Venetoclax, a BCL-2 inhibitor, to standard high dose therapy prior to autologous stem cell transplant (ASCT).
  Venetoclax is a novel, orally bioavailable, small-molecule B-cell lymphoma-2 (Bcl-2) family inhibitor.

SUMMARY:
The purpose of this study is to determine the correct dose and safety of adding a new cancer drug, Venetoclax, to a standard combination of chemotherapy drugs used prior to Autologous stem cell transplant (ASCT) in participants with Non-Hodgkin Lymphoma (NHL). In this study, Venetoclax will be added to BEAM (BCNU or carmustine, etoposide, cytarabine or ara-c, and melphalan). All NHL participants are admitted for conditioning chemotherapy which is given prior to the infusion of stem cells.

Venetoclax is a new anti-cancer drug that works by targeting a protein (known as the Bcl-2 protein). By inhibiting or "blocking" this protein, a downstream cascade occurs which results in cancer cells to die. Adding Venetoclax to the standard BEAM conditioning chemotherapy with autologous stem cell transplant is believed to increase the chance of remission. Venetoclax is Food and Drug Administration (FDA) approved for participants with chronic lymphocytic leukemia (CLL). However, Venetoclax is investigational for this study because it is not yet approved for use in participants with NHL or in combination with BEAM chemotherapy.

DETAILED DESCRIPTION:
The primary objective of this study is to establish the safety of V-BEAM conditioning regimen prior to autologous stem cell transplant in order to identify the recommended phase II dose (RPD2). This study will also seek to compare time to neutrophil engraftment and time to platelet engraftment of participants who receive V-BEAM and ASCT, compared to historical controls and among cohorts. And finally, it will determine the Progression Free Survival (PFS) and Overall Survival (OS) of V+BEAM followed by ASCT relative to historical controls of BEAM alone followed by ASCT.

This will be a single-institution, open label, phase I study designed to evaluate the safety of this combination. The target population will be participants with NHL who are eligible for ASCT. Dose escalation will proceed using a standard 3 + 3 design with 5 dose levels, a minimum of 6 participants and a maximum of 30 participants will be required to identify the RP2D. If a participant does not take all scheduled doses of Venetoclax according to his/her cohort, the participant will be replaced because he/she has not taken enough drug to confirm safety at that dose level.

Once the conditioning regimen has been delivered and autologous stem cells have been infused there is no further disease-directed treatment as part of this protocol. In accordance with routine practice the bone marrow transplant program at the Cleveland Clinic, participants receive supportive care and follow-up until disease relapse or death. In the absence of treatment delays during the conditioning regimen due to adverse events, participants will remain on study for 24 months or until one of the following criteria applies:

* Disease progression
* Intercurrent illness that prevents further administration of treatment
* The investigator considers it, for safety reasons, to be in the best interest of the participant.
* General or specific changes in the participant's condition rendering the participant unacceptable for further treatment in the judgment of the investigator.
* Participants decision to withdraw from treatment (partial consent) or from the study (full consent)
* Pregnancy during the course of the study for a child-bearing participant
* Death, or
* Sponsor reserves the right to temporarily suspend or prematurely discontinue this study.

Participants will be followed for toxicity for 24 months after hospital discharge or until a protocol approved outcome. The first 3 months will be at the treating center and continued recommended follow-up should be at a minimum of 6 months, 12 months, 18 months and 24 months after hospital discharge or as clinically appropriate according to local practices.

The clinical course of each event will be followed until resolution, stabilization, or until it has been determined that the study treatment or participation is not the cause.

Serious adverse events that are still ongoing at the end of the study period will necessitate follow-up to determine the final outcome. Any serious adverse event that occurs after the study period and is considered to be possibly related to the study treatment or study participation will be recorded and reported immediately.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed Non-Hodgkin Lymphoma (NHL) including T-cell lymphomas, after at least one prior systemic treatment regimen such as CHOP, R-CHOP, CHOEP, R-EPOCH, R-HyperCVAD, BR, VR-CAP alternating with rituximab and cytarabine, etc.
* Patients in complete or partial remission, or in the case of patients with stable or refractory disease are undergoing autologous transplantation because it has been recommended by their treating physician as representing their best treatment option.
* ECOG Performance status ≤ 2 at time of consent [See Appendix I].
* Patients must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 8.0 g/dl
  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelet count ≥ 75,000/mcL
  * Total bilirubin ≤ 1.5X the upper limit of normal (ULN) unless a known history of impaired bilirubin conjugation such as Gilbert's.
  * AST (SGOT) ≤ 2.5 X institutional ULN
  * ALT (SGPT) ≤ 2.5 X institutional ULN
  * Patients must have a calculated serum creatinine clearance > 50 mL/min using Cockcroft-Gault calculation or based on 24-hour urine collection performed within 7 days prior to treatment.
  * Cardiac ejection fraction >45% or clearance by PI or Cardiology
  * DLCO of >45% predicted or clearance by PI or Pulmonology
* Specific guidelines will be followed regarding inclusion of NHL based on Hepatitis B serological testing as follows:

  * HBsAg negative, HBcAb negative, HBsAb negative patients are eligible.
  * HBsAg negative, HBcAb negative, HBsAb positive patients are eligible.
  * Patients who test positive for HBsAg are ineligible.
  * Patients with HBsAg negative, but HBcAb positive (regardless of HBsAb status) should have a HBV DNA testing performed and protocol eligibility determined as follows:

    * If HBV DNA is positive, the patient is ineligible.
    * If HBV DNA is negative, the patient may be included but must undergo HBV DNA PCR testing monthly x 3 months beginning from the start of treatment
* Female patients who are not surgically sterile or postmenopausal (for at least 1year) must practice at least one of the following methods of birth control throughout the duration of study participation and for at least 30 days after study treatment:

  * Total abstinence from sexual intercourse
  * A vasectomized partner
  * Hormonal contraceptives (oral, parenteral, vaginal ring, or transdermal) that started at least 3months prior to study drug administration
  * Double-barrier method (condom+diaphragm or cervical cup with spermicidal contraceptive sponge, jellies, or cream)
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria: The presence of any of the following will exclude a patient from study enrollment:

* Patients who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Prior treatment toxicities have not resolved to ≤ Grade 2 according to NCI CTCAE Version 5.0 (except clinically unrelated toxicities such as alopecia or peripheral neuropathy).
* Patients receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Venetoclax or other agents used in this study.
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who are pregnant or breastfeeding will be excluded from this study because carmustine, etoposide, cytarabine, and melphalan are chemotherapeutic agents with the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with carmustine, etoposide, cytarabine, and melphalan, breastfeeding should be discontinued if the mother is treated with these agents. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Venetoclax. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated. HIV testing prior to enrollment is not required for screening but strongly encouraged for patients with no documented prior HIV assessment.
* Malabsorption syndrome or other condition that precludes enteral route of Venetoclax administration
* Patients with metastatic solid tumor malignancies. Patients who have early stage solid tumors and have completed curative treatment are eligible at the discretion of the primary investigator. Patients with unresected but localized stage prostate cancer or other carcinomas in situ that are undergoing observation are also allowed. Patients with transformed lymphoma and/or underlying indolent lymphoproliferative disorder are allowed at the discretion of the investigator.
* Major surgery, other than diagnostic surgery, within 2 weeks.
* Medical condition requiring chronic use of high dose systemic corticosteroids (i.e., doses of prednisone higher than 10 mg/day or equivalent). Brief (<15 days) treatment with glucocorticoids (prednisone 100 mg by mouth daily, or equivalent) is acceptable.
* Patients with chronic use of moderate or strong CYP3A4 modulators (inhibitor or inducer) or use of a P-gp inhibitor, or a P-gp substrate with a narrow therapeutic index are prohibited. A washout period of 7 days is required prior to Venetoclax dosing if a prohibited medication is discontinued. Lists including medications or substances known or with the potential to interact with the specific CYP3A4 isoenzymes and P-gp are provided in Appendix II.
* Concomitant medications that fall into the categories below could potentially lead to adverse reactions and should be considered cautionary (except where noted). Medications and cautionary medications that fall into the categories within this section can be found at http://medicine.iupui.edu/clinpharm/ddis/main-table. If a potential study patient is taking any of the medications in the categories described below, the investigator will assess and document the use of medications known or suspected to fall in the following medication categories:

  * Moderate/Weak CYP3A inducers such as efavirenz and oxcarbazepine.
  * CYP2C8 substrates such as thiazolidinediones (glitazones) and select statins (because of expected inhibition of the metabolism of CYP2C8 substrates by Venetoclax).
  * CYP2C9 substrates such as tolbutamide (because of expected inhibition of the metabolism of CYP2C9 substrates by Venetoclax). It is recommended to exclude CYP2C9 substrates with a narrow therapeutic index such as phenytoin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety of intervention as defined by hematopoietic non-engraftment (failure of either ANC engraftment or platelet engraftment). | Up to 30 days after Autologous Stem Cell Transplant (ASCT)
  Safety of intervention will be measured by the effect on hematologic engraftment (engraftment Dose Limiting Toxicity DLT). This includes failure of absolute neutrophil count (ANC) engraftment OR platelet engraftment.
  • Failure of ANC engraftment which is defined as failure to engraft by day 15.
  OR
  • Failure of platelet engraftment which is defined as failure to engraft by day 30.

SECONDARY OUTCOMES:
Time to neutrophil engraftment | 24 months after hospital discharge
  Compare time to neutrophil engraftment of patients who receive V-BEAM followed by ASCT, compared to historical controls and among cohorts.
Time to platelet engraftment | 24 months after hospital discharge
  Compare time to platelet engraftment of patients who receive V-BEAM followed by ASCT, compared to historical controls and among cohort.
Progression-free survival (PFS) | 24 months after hospital discharge
  Determine the Progression Free Survival (PFS) of V+BEAM followed by ASCT relative to historical controls of BEAM alone followed by ASCT.
  PFS is defined as the time from entry onto study until lymphoma progression or death from any cause. PFS reflects tumor growth and, therefore, occurs prior to the endpoint of overall survival.
Overall Survival (OS) | 24 months after hospital discharge
  Determine the Overall Survival (OS) of V+BEAM followed by ASCT relative to historical controls of BEAM alone followed by ASCT.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Winter, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio